CLINICAL TRIAL: NCT03974243
Title: Phase Ib/IIa Study of Chiauranib in Combination With Chidamide in Patients With Relapsed/Refractory Non-Hodgkin's Lymphoma
Brief Title: Chiauranib in Combination With Chidamide in Patients With Relapsed/Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR106
Record Dates: First submitted 2019-05-30; First posted 2019-06-04 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2021-08

CONDITIONS: Non-hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — chiauranib; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): In this arm, patients would be given the regimen composed of Chiauranib and Chidamide orally.
  Intervention: Drug: Chiauranib and Chidamide
  Interventions: Drug: Chiauranib; Drug: Chidamide

INTERVENTIONS:
Drug: Chiauranib — In the lead-in period, patients take 50mg Chiauranib capsules on the forth day .
  In the subsequent treatment cycles, Chiauranib capsules are given orally once daily, 28 days as a cycle.
  Other Names: CS2164
Drug: Chidamide — In the lead-in period, patients take a single dose of Chidamide tablet on the first day and then off for 3 days before the first cycle begins. In the subsequent treatment cycles, Chidamide tablets are given orally on Day 1,4,8,11,15,18,22 and 25 of each cycle. 28 days as a cycle
  Other Names: CS055

SUMMARY:
The purpose of this dose-escalation study is to assess the safety and tolerability of treatment with Chiauranib and Chidamide administered orally over a range of doses in patients with relapsed or refractory non-Hodgkin's lymphoma, in the meantime, exploring the pharmacodynamic profile and latent biomarkers accompany with Chiauranib and Chidamide , as well as the relevancy of which and clinical benefit.

DETAILED DESCRIPTION:
The purpose of this study is to assess the tolerability and safety include adverse events, vital signs, laboratory tests ,etc., of a range of doses of Chiauranib and Chidamide in patients with relapsed or refractory non-Hodgkin's lymphoma, and to determine the dose limit toxicity and the maximum tolerable dose.

In the meantime, exploring the pharmacodynamic profile and latent biomarkers accompany with Chiauranib and Chidamide , as well as the relevancy of which and clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, aged ≥ 18 yrs and ≤70 yrs;
2. Patients with NHL refractory to at least 2 different chemotherapies , for which no standard therapy exists;
3. At least 1 lesion can be accurately measured, as defined by Lugano 2014 criteria.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
5. Subjects received anti-cancer therapy (including chemotherapy, radiotherapy, immunotherapy and surgical therapy, et al) should beyond 4 weeks prior to study entry; Subjects received mitomycin chemotherapy should beyond 6 weeks prior to study entry; Subjects received autologous stem cell transplantation should beyond 3 months prior to study entry;
6. Laboratory criteria are as follows:

   Complete blood count: hemoglobin (Hb) ≥90g/L ; absolute neutrophil count (ANC) ≥1.5×109/L ; platelets >=90×109/L Biochemistry test: total bilirubin≦1.5×ULN; alanine aminotransferase(ALT) ,aspartate aminotransferase(AST)≦1.5×ULN; (ALT,AST≦5×ULN if liver involved) ;serum creatinine(cr)≦1.5×ULN; Coagulation test: International Normalized Ratio (INR) < 1.5
7. Life expectancy of at least 3 months.
8. Willingness to sign a written informed consent document.

Exclusion Criteria:

1. Clinical evidence of central nervous system involvement
2. Patients with prior invasive malignancies with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or cervical carcinoma in situ, unless received curative treatment and with documented evidence of no recurrence in the past five years;
3. Previous treatment with HDAC inhibitors(include Chidamide) or aurora kinase(include Chiauranib) inhibitors;
4. Have uncontrolled or significant cardiovascular disease, including:

   1. Congestive heart failure, unstable angina pectoris, myocardial infarction within 6 months prior to study entry; arrhythmia, or Left Ventricular Ejection Fraction (LVEF) < 50% requiring treatment with agents during screening stage.
   2. primary cardiomyopathy(dilated cardiomyopathy, hypertrophic cardiomyocyte, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, et,al)
   3. History of significant QT interval prolongation, or Corrected QT Interval (QTc) > 450 ms prior to study entry
   4. Symptomatic coronary heart disease requiring treatment with agents
   5. Uncontrolled hypertension (> 140/90 mmHg) by single agent;
5. Have active bleeding current thrombotic disease, patients with bleeding potential ,or receiving anticoagulation therapy; within 2 months prior to screening;
6. Proteinuria positive(≥1g/24h);
7. History of deep vein thrombosis or pulmonary embolism;
8. Have unsolved toxicities (> grade 1) from prior anti-cancer therapy;
9. Have clinical significant gastrointestinal abnormality, e.g., unable to swallow, chronic diarrhea, ileus, that would impair the ingestion,transportation or absorption of oral agents, or patients undergone gastrectomy;
10. History of organ transplantation ，Allogeneic bone marrow transplantation or autologous stem cell transplantation;
11. High-risk surgery for vital organs within 6 weeks prior to screening or the investigators determined that other surgical wounds did not heal well;
12. Serologically positive for HIV, hepatitis B or C, or other serious infectious diseases;
13. History of interstitial lung disease(ILD);
14. Any mental or cognitive disorder, that would impair the ability to understand the informed consent document or the operation and compliance of study;
15. Candidate with drug and alcohol abuse;
16. Participants of reproductive potential not willing to use adequate contraceptive measures for the duration of the study (both male and female participants).Pregnant or breastfeeding women. Female participants must have a negative urinary or serum pregnancy test when done or have evidence of post-menopausal status (Defined as absence of menstruation for greater than 12 months, bilateral oophorectomy or hysterectomy);
17. Any other condition which is inappropriate for the study in the opinion of the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
dose-limiting toxicity (DLT) | Day 1 - 28

SECONDARY OUTCOMES:
Area under the concentration versus time curve (AUC) | Day 1 of the lead-in period and Day 1 of the combination therapy
  pharmacokinetic profile of Chiauranib in combination with Chidamide
Peak plasma concentration (Cmax) | Day 1 of the lead-in period and Day 1 of the combination therapy
  pharmacokinetic profile of Chiauranib in combination with Chidamide
Time of Cmax (Tmax) | Day 1 of the lead-in period and Day 1 of the combination therapy
  pharmacokinetic profile of Chiauranib in combination with Chidamide
Objective response rate | About 21 weeks
complete response rate | About 21 weeks
disease control rate | About 21 weeks
time to progression | About 21 weeks
  duration from date of treatment until the date of first documented progression
Progression free survival | About 21 weeks
  From date of treatment until the date of first documented progression or date of death from any cause, whichever came first
Duration of response | About 21 weeks
  From the first date of response until the date of first documented progression
Adverse events | About 21 weeks
  Number of participants with treatment-related adverse events according to CTCAE V4.03
Any single mutation of oncogene and copy number variation in ctDNA(single gene analysis) | day -1 of therapy
Mutation of polygene and copy number variation in signal pathway(multi-gene analysis) | day -1 of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided